CLINICAL TRIAL: NCT02750358
Title: Feasibility Study of Adjuvant Enzalutamide for the Treatment of Early Stage AR(+) Triple Negative Breast Cancer
Brief Title: Feasibility Study of Adjuvant Enzalutamide for the Treatment of Early Stage AR (+) Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Medivation, Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-307
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Early Stage; Triple Negative Breast Cancer
Keywords: Enzalutamide; 15-307
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — enzalutamide; Restraint, Physical; Weights and Measures

ARMS (1):
- Enzalutamide (Experimental): 160mg orally as daily continuous dosing for 52 weeks. Patients will be seen for protocol visits every 4 weeks (+/- 2 week window) for the first 12 weeks followed by every 12 weeks (+/- 2 week window) to complete 52 weeks. An assessment will also be performed at 52 weeks (+ 4 week window).
  Interventions: Drug: Enzalutamide; Behavioral: assessment

INTERVENTIONS:
Drug: Enzalutamide
Behavioral: assessment
  Other Names: Functional Assessment of Cancer Therapy-Breast (FACT-B) scale

SUMMARY:
This trial is designed to determine the feasibility of 1 year of adjuvant enzalutamide, an androgen receptor (AR) antagonist for the treatment of patients with early stage, AR(+) triple negative breast cancer (TNBC).

ELIGIBILITY:
The study population for Step 1 must meet the following eligibility criteria:

Inclusion Criteria:

* Stage 1, 2 or 3 invasive breast cancer which is triple negative. Triple negative breast cancer is defined as ER <1, PR <1 and HER2 0 or 1+ or FISH not amplified if IHC 2+.
* AR testing may be performed while patient is undergoing other adjuvant therapy (i.e., surgery, chemotherapy, radiation).
* Willing and able to provide informed consent. Woman at least 18 years of age.
* Patient is a candidate for treatment of their early stage breast cancer.

The study population for Step 2 will meet the eligibility criteria:

Inclusion Criteria:

* Stage 1, 2 or 3 invasive breast cancer which is triple negative. Triple negative breast cancer is defined as ER <1%, PR <1% and HER2 0 or 1+ or FISH not amplified if IHC 2+.
* AR(+), defined as ≥1% nuclear staining by IHC testing. The assessment of AR expression may have been performed any time in the past and is not limited to participation in Step 1.
* Any neoadjuvant or adjuvant chemotherapy regimen is permitted. Prior chemotherapy for the treatment of this breast cancer is not required.
* At least 4 weeks from end of surgery, chemotherapy, or radiotherapy with resolution of any toxicity to Grade 1 or less, excluding alopecia.
* Patients are eligible to participate within 6 months of completion of therapy for their breast cancer. This includes prior radiation therapy if needed.
* ECOG performance status of 0 or 1.
* Willing and able to provide informed consent.
* Woman at least 18 years of age.
* Able to swallow study drug and comply with study requirements.
* Women of childbearing potential must have a negative pregnancy test and must agree to use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration.
* Is not breastfeeding at screening and will not breastfeed throughout the study period and for at least 3 months after final drug administration.

Exclusion Criteria:

Each patient eligible to participate in this study must NOT meet any of the following exclusion criteria.

* Any severe concurrent disease, infection or comorbid condition that renders the patient inappropriate for enrollment in the opinion of the investigator or interferes with the patient's ability to participate in the study requirements.
* Evidence of metastatic/Stage 4 breast cancer
* History of another invasive cancer within 5 years with the exceptions of nonmelanoma skin cancers and AJCC Stage 0 or 1 cancers that have a remote probability of recurrence in the opinion of the investigator
* Absolute neutrophil count < 1500/μL, platelet count < 75,000/μL, or hemoglobin < 9 g/dL (5.6 mmol/L).
* Total bilirubin > 1.5 times upper limit of normal (ULN) unless an alternate nonmalignant etiology exists (eg, Gilbert's disease). Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times ULN.
* Creatinine > 1.5 times ULN or an estimated creatinine clearance < 50 mL/minute calculated using the Cockcroft-Gault equation.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past. Also, history of loss of consciousness or transient ischemic attack within 12 months before day 1
* An active gastrointestinal disorder affecting absorption (eg, gastrectomy, active peptic ulcer disease, uncontrolled celiac)
* Hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole and butylated hydroxytoluene.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05-19; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The treatment discontinuation rate of enzalutamide in the adherent population | 3 years
  feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Kings County Hopsital Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Woodhull Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Queens Hospital Center, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/